CLINICAL TRIAL: NCT04996888
Title: A Prospective Multicenter Study on the Effect of Preoperative Automatic Reminder System on Colonoscopy
Brief Title: Effect of Preoperative Automatic Reminder System on Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EA-21-007
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Colonoscopy
Keywords: the quality of bowel preparation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with AI preoperative automatic reminder system (Experimental): After receiving regular instructions at the time of their appointment to discuss colonoscopy and education about colonoscopy provided by one nurse, including the importance of bowel preparation, the side effects of the agents used, and the exact preparation instructions, the patients in the experimental group will be sent a message and a phone call by AI system on the day before colonoscopy, which will emphasize the importance of bowel preparation, the directions for use and side effects of purgatives, the proper food type, and the start time.
  Interventions: Device: AI based preoperative automatic reminder system
- without AI preoperative automatic reminder system (No Intervention): The patients in the control group accept colonoscopy routinely without AI based preoperative automatic reminder system. All patients will receive regular instructions at the time of their appointment to discuss colonoscopy and education about colonoscopy provided by one nurse, including the importance of bowel preparation, the side effects of the agents used, and the exact preparation instructions.

INTERVENTIONS:
Device: AI based preoperative automatic reminder system — the patients in the experimental group will be sent a message and a phone call by AI system on the day before colonoscopy, which will emphasize the importance of bowel preparation, the directions for use and side effects of purgatives, the proper food type, and the start time. The system is an non-invasive AI system.
  Arms: with AI preoperative automatic reminder system

SUMMARY:
In this study, the investigators proposed an artificial intelligence-based preoperative automatic reminder system on colonocopy, which can improve the quality of bowel preparation and the rate of polyps and adenomas detection.

DETAILED DESCRIPTION:
Despite advances in bowel preparation methods, bowel preparation is inadequate in up to one-third of all colonoscopies in reported series. Inadequate bowel cleansing results in negative con-sequences for the examination, including incomplete visualization of the colon, missed lesions(22-48%), procedural difficulties, prolonged procedure time and reduced time interval until follow-up, and an estimated 12-22% increase in overall colonoscopy cost.

The adequacy of a bowel preparation is closely linked to patient compliance with both dietary and purge instructions. Previous work has shown that 18-23.5% of the patients with poor preparation had failed to follow preparation instructions. One study performed in Asia showed that non-compliance with bowel preparation instructions, lower education level, and a long wait for the colonoscopy appointment were independent risk factors for poor bowel preparation. A survey among doctors showed that gastroenterologists with the highest number of patients with inadequate bowel preparation believed that patients are unwilling to follow preparation instructions, struggle with the prescribed diet, and are unable to tolerate the full course of purgative. It is reasonable to hypothesis that efforts to improve education and maximize patient compliance during the preparatory period will enhance the efficacy of bowel preparation.

A research has shown that telephone-based re-education about the details of bowel preparation on the day before colonoscopy significantly improved the quality of bowel preparation and polys detection rate. In recent years, artificial intelligence (AI) has been successfully applied in multiple medical fields. But there has not been an artificial-intelligence-based system which can automatically remind patients of the details of bowel preparation on the day before colonoscopy.

In this study, we proposed an artificial intelligence-based preoperative automatic reminder system on colonoscopy, which can improve the quality of bowel preparation and the rate of polyps and adenomas detection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 50-75 years old;
2. Able to read, understand and sign informed consent
3. The investigator believes that the subjects can understand the process of the clinical study, are willing and able to complete all study procedures and follow-up visits, and cooperate with the study procedures
4. Outpatients requiring colonoscopy

Exclusion Criteria:

1. colorectal surgical history
2. Severe colonic stricture or obstructive tumor
3. Obvious gastroparesis or gastric outlet obstruction or intestinal infarction
4. Pregnant or lactating women
5. Dysphagia or impaired swallowing reflex or mental state
6. Intestinal obstruction or perforation is known
7. Severe chronic renal failure（CCR< 30ml/min）
8. Severe congestive heart failure（NYHA ⅢorⅣ）
9. Uncontrolled hypertension( systolic pressure>170mmHg，diastolic pressure>100mmHg)
10. Dehydration or electrolyte disorder
11. Toxic colitis or megacolon
12. Inable to give informed consent
13. Hemodynamic instability

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Estimated)
Dates: Start 2021-08-04 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
the rate of adequate bowel preparation | From the beginning to the end of colonoscopy
  The numerator is the number of patients qualified for intestinal preparation, and the denominator is the number of all patients undergoing colonoscopy. The definition of intestinal preparation qualification is: e-bbps qualification is defined as colonoscopy with e-bbps ≥ 6; BBPS is defined as enteroscopy with scores ≥2 for ascending colon, transverse colon and descending colon. At the same time, if one or more of the following conditions are met, intestinal preparation is considered insufficient: (1) colonoscopy with e-bbps <6 is insufficient（ 2) Cancel colonoscopy due to poor intestinal preparation or personal reasons（ 3) Incomplete colonoscopy.

SECONDARY OUTCOMES:
Detection rate of adenoma | A month
  The numerator is the number of patients diagnosed with adenomas, and the denominator is the total number of patients undergoing colonoscopy.

OTHER OUTCOMES:
Detection rate of polyp | A month
  The numerator is the number of patients diagnosed with polyp, and the denominator is the total number of patients undergoing colonoscopy.
Rate of willing to repeat intestinal preparation | Six month
  the numerator is the number of patients who are willing to prepare for colonoscopy again after inquiry due to timely treatment in the future or insufficient intestinal preparation, and the denominator is the number of patients who receive colonoscopy
Instructions compliance analysis | From the beginning to the end of colonoscopy
  Failure to comply with intestinal preparation is defined as failure to take laxatives on time, failure to comply with dietary restrictions, and acknowledgement of failure to comply with instructions, including insufficient dosage of intestinal preparation solution, insufficient duration of completion of intestinal preparation solution, and insufficient hydration
Attendance rate | From the beginning to the end of colonoscopy
  the numerator is the number of patients on time, and the denominator is the number of patients undergoing enteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yu W Honggang, Doctor, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin hospital of Wuhan University, Wuhan, Hubei, China